CLINICAL TRIAL: NCT01105299
Title: Bioequivalence Study of CJ Anastrozole 1mg Tablet and Arimidex® 1 mg Tablet
Brief Title: Bioequivalence Study of Anastrozole 1 mg Tablet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Hyeong-Seok Lim/associate professor, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_ANS_B01
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: bioequivalence; anastrozole; Healthy subjects; Antineoplastic Agents; Therapeutic Uses; Enzyme Inhibitors
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CJ anastrozole 1 mg tablet

SUMMARY:
The purpose of this study is to characterize and compare the bioequivalence of CJ anastrozole [CJ Cheiljedang corp., Seoul, Korea] with Arimidex® [AstraZeneca, Wilmington, DE, USA].

DETAILED DESCRIPTION:
This study was conducted to characterize and compare the pharmacokinetic and safety profiles and the bioequivalence of a newly developed new generation aromatase inhibitor (CJ anastrozole) with existing anastrozole formulation (Arimidex®) in healthy Korean volunteers. This study is designed as single-dose, randomized, double-blind, 2-way crossover trial. Participants were randomized to receive 1 mg of either the CJ anastrozole or Arimidex, followed by a 3-week washout period. And then the alternate formulation was administered. After 10-hour overnight fast drug was administered. For analysis of pharmacokinetic properties, including Cmax and AUClast, blood samples were obtained at 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, and 216 hours after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers in the age between 19 to 55 years old
* Subjects were neither congenital nor chronic diseases.
* Subjects were selected after passing a clinical screening procedure that included a physical examination and laboratory tests.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.

Exclusion Criteria:

* Any history of a clinical condition which might affect drug absorption, distribution, metabolism or excretion or might be risk factors, e.g. clinically significant disorder in heart, liver, respiratory system, liver, kidney, gastrointestinal system and CNS
* Had a history of myocardial infarction, stroke, hypertension, arrhythmia, coronary artery disease, disease of neuropsychiatry, gastrointestinal system surgery (excluding appendectomy, herniotomy)
* Current clinically significant disorder in history taking or physical examination
* Acute disease within 14 days preceding the first application of study medication
* Had an relevant allergic disease
* Had history of hypersensitivity to drugs or any food
* Positive for Hepatitis B antigen, Hepatitis C antibody, HIV antibody, or High Quality Syphilis Reagin Test
* Excessive caffeine, alcohol intake and smoker(caffeine>5 units/day, alcohol>3 units/day(1 unit = pure alcohol 10ml), cigarettes> 20 cigarettes /day)
* Subjects who excessive alcohol intake or drug which affect drug metabolism enzyme intake within 30 days preceding study
* History of drug abuse or positive for urinary testing of drugs abuse (amphetamine, barbiturates, cocaine, opioids, benzodiazepines etc.)
* Has donated whole blood within 60days or apheresis within 14days preceding the first application of study medication
* Received other investigational drug within 60days preceding the first application of study medication
* Taken any herbal medicine within 30days, prescription medication within 14 days or over-the-counter drug (except for vitamins, minerals) within 10days preceding the first application of study medication (might affect this study or safety of subjects as judged by the investigator)
* Subjects could not eat ASAN MEDICAL CENTER standard meal or were unsuitable for this study as judged by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, MD, Principal Investigator — Asan Medical Center

REFERENCES:
- [Derived] Noh YH, Ko YJ, Cho SH, Ghim JL, Choe S, Jung JA, Kim UJ, Jin SJ, Park HJ, Song GS, Lim HS, Bae KS. Pharmacokinetic comparison of 2 formulations of anastrozole (1 mg) in healthy Korean male volunteers: a randomized, single-dose, 2-period, 2-sequence, crossover study. Clin Ther. 2012 Feb;34(2):305-13. doi: 10.1016/j.clinthera.2012.01.008. Epub 2012 Jan 26. PMID 22281018
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks